CLINICAL TRIAL: NCT04624867
Title: A Phase I Study to Assess Skin Irritation and Sensitization of HP-1050 Transdermal System Compared to XULANE in Healthy Adult Females
Brief Title: Study Will Assess Skin Irritation and Sensitization for HP-1050 Patch
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Noven Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-1050-US-02
Record Dates: First submitted 2020-10-22; First posted 2020-11-12 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cumulative Irritation and Sensitization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HP-1050 patch (Experimental): HP-1050 and Xulane will be administered simultaneously.
  Interventions: Drug: HP-1050 Patch

INTERVENTIONS:
Drug: HP-1050 Patch — Both articles, HP-1050 and XULANE patch, will be applied simultaneously on the back of each subject.

SUMMARY:
A randomized, evaluator-blinded study to assess skin irritation and skin sensitization of HP-1050 transdermal system (HP-1050) in comparison to XULANE patch in healthy female volunteers.

DETAILED DESCRIPTION:
This is a dual-center, evaluator-blinded, randomized phase 1 study evaluating skin irritation and skin sensitization of HP-1050 transdermal system in comparison to XULANE patch in healthy female volunteers. The study will consist of a 4-week Screening Phase and a Treatment Phase. The Treatment Phase will consist of the following periods: an Induction Period, a Rest Period followed by a Challenge Period and if needed, a Re-Challenge Period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant, non-lactating females 18-35 years of age (inclusive0 and who are candidates for hormonal contraception;
* Subjects who have previously used hormonal contraceptives without complications or naïve subjects for whom hormonal contraceptives are not contraindicated in the opinion of the Principal Investigator;
* Subjects who are willing to stop using any current contraceptives for the duration of the study;

Exclusion Criteria:

* Subjects who are currently taking or have taken oral hormonal contraceptives within 30 days prior to the first patch application;
* Subjects who are currently using any long-acting hormonal method of contraception or has used them within the past 3 months;
* Subjects who have a contraindication for estrogen or norelgestromin, or subjects who have a history of sensitivity to estrogen or norelgestromin or any related derivatives;

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Skin Irritation Evaluation | 21 days
  To evaluate skin irritation after exposure to HP-1050 compared to XULANE®
Sensitization Evaluation | 48 hours
  To evaluate skin sensitization after exposure to HP-1050 compared to XULANE®

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Missouri, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided